CLINICAL TRIAL: NCT03349502
Title: Pilot Study of Safety and Efficacy of Lymphodepletion Followed by MG4101 Administered Intravenously to Patients With Refractory or Relapsed AML
Brief Title: MG4101 for Refractory or Relapsed AML
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Seoul National University Hospital (Other)
Responsible Party: Principal Investigator, YOUNGIL KOH, Assistant Professor, Seoul National University Hospital
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: H-1705-065-853
Record Dates: First submitted 2017-11-17; First posted 2017-11-21 (Actual); Last update posted 2023-04-18 (Actual); Status verified 2023-04

CONDITIONS: Acute Myeloid Leukemia
Keywords: Allogeneic natural killer cell, MG4101
MeSH Terms: conditions — Leukemia, Myeloid, Acute

STUDY DESIGN:
Intervention Model Description: Single center, single arm, open-labeled phase 2 trial
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- MG4101 (Experimental): MG4101 administration (Not yet commercialized)
  1. Dosage Bwt<50 : 2.0 x109 cells (2 bags) 50≤Bwt<70 : 3.0 x109 cells (3 bags) 70≤Bwt<100 : 4.0 x109 cells (4 bags) Bwt≥100 : 5.0 x109 cells (5 bags)
  2. Duration and frequency
     * Intravenous over 1 hour
     * Day 4, Day 11, Day 18 of each cycle
  Interventions: Drug: MG4101

INTERVENTIONS:
Drug: MG4101 — Administration of study drug (MG4101) for the patients with refractory or relapsed acute myeloid leukemia (Single arm)
  Other Names: Allogeneic natural killer cell

SUMMARY:
This study is a single center, single arm, open-labeled phase 2 clinical study. The aim of this study is to investigate the efficacy and safety of allogeneic natural killer cell (MG4101). After lymphodepletion with fludarabine and cyclophosphamide, the patient will receive MG4101. Each cycle consists of 28 days, and a total of 2 cycles of MG4101 will be administered with IL-2 to activate the study drug. The efficacy of MG4101 will be evaluated after 8 weeks from the first day of treatment. We will evaluate the safety of the drug measuring the vital sign, laboratory tests, and adverse events.

DETAILED DESCRIPTION:
Acute myeloid leukemia is a hematologic malignancy of myeloid lines leukocyte. In Korea, acute leukemia accounts for 87% of all leukemia and the incidence of acute myeloid leukemia is twice as high as acute lymphoblastic leukemia. The general treatment strategy for AML has not changed over the past 30 years. In adult AML, about 70 to 80% of the patients achieve complete remission after the intensive induction chemotherapy, but disease recurrence is relatively common. After the recurrence, the patients with good physical condition receive intensive salvage chemotherapy followed by allogeneic hematopoietic stem cell transplantation. But even with the intensive treatment, the long-term survival rate is only about 25%.

MG4101 is the natural killer (NK) cell product that is activated in vitro after obtaining through leukapheresis from a healthy donor. The allogeneic NK cell is well known to have anti-leukemic effect in allogeneic stem cell transplantation. As it is widely reported that the lymphodepletion is essential in adoptive cell transfer therapy, MG4101 will be administered after the conditioning with cyclophosphamide and fludarabine. And after the infusion of MG4101, IL-2 will be infused together to activate the study drug.

In the dose-finding phase 1 study of MG4101 (NCT01212341), the maximal tolerated dose was estimated to exceed 3x10^7 cells/kg. The patients will receive 2.0x10^9 to 5.0x10^6 cells in each cycle, based on the weight.

The protocol is as follows:

Cyclophosphamide and fludarabine will be administered at the dose of 250 mg/m2/day and 20 mg/m2/day, respectively, for 3 days from the start of the treatment. On the 4th, 11th and 18th day, the study drug, MG4101, will be administered intravenously, followed by 3 days of IL-2. The response will be assessed on the 28th, 56th and 112th day. The adverse event will be observed for 56 days after the initiation of the treatment.

ELIGIBILITY:
Inclusion Criteria:

* Age between 18 to 65
* Eastern Cooperative Oncology Group (ECOG) performance status 0,1,2
* Informed consent
* Diagnosed with acute myeloid leukemia by 2016 WHO criteria
* Failure to achieve complete remission after the second line of standard chemotherapy
* Relapse after the second line of standard chemotherapy and not eligible for the allogeneic stem cell transplantation
* Adequate major organ function

Exclusion Criteria:

* Acute promyelocytic leukemia
* Central nervous system involvement of the leukemia
* Hypersensitivity to IL-2
* Previous cell therapy
* Impaired major organ function

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2017-11-01 (Actual); Primary Completion 2020-03-30 (Actual); Study Completion 2020-04-30 (Actual)

PRIMARY OUTCOMES:
Overall response rate | After completion of 2 cycles of treatment (Day 56 from the initiation of the treatment)
  Sum of complete remission (less than 5% of blast in normocellular or hypercellular bone marrow, no remnant leukemic cell or chloroma, absolute neutrophile count more than 1x10^9/L, platelet count more than 100x10^9/L) and complete remission with incomplete blood count recovery (less than 5% of blast in normocellular or hypercellular bone marrow with acute neutrophil count less than 1x10^9/L or platelet count less than 100x10^9/L)

SECONDARY OUTCOMES:
Overall survival | At the end of the study (Day 112 from the initiation of the treatment)
  From the initiation of the study to the death of any cause or censoring
Duration of complete remission | At the end of the study treatment (Day 112 from the initiation of the treatment)
  Cumulative incidence of relapse

CONTACTS AND LOCATIONS:
Overall Officials: Youngil Koh, MD, Principal Investigator — Seoul National University Hospital
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

IPD SHARING:
Plan to Share IPD: No
There is no plan to make individual participant data